CLINICAL TRIAL: NCT00672711
Title: Susceptibility to Chronic Post-Traumatic Extremity Pain
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Collaborators: Beaumont Foundation of America (Other); Oakland University (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-200
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
Keywords: Complex Regional Pain Syndrome; Chronic Post-surgical Pain; Genetic susceptibility; COMT
MeSH Terms: conditions — Chronic Pain; Complex Regional Pain Syndromes; Pain, Postoperative; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- C: APS
- B: HPS
- A: LPS

SUMMARY:
The association between the COMT haplotypes and the presence or absence of CPSP or CRPS will be assessed stratifying the patients based on the individual categories of trauma or elective surgery.

DETAILED DESCRIPTION:
This will be a prospective association study in which we will recruit patients who have experienced single extremity trauma, or who have scheduled elective surgery on a single extremity. HRQoL will be determined at recruitment. We will identify their haplotypes and genotypes for 4 linked SNPs in the coding region of COMT as described by Diatchenko [2]. Patients will receive follow-up at 3 and 6 months following trauma or surgery. Individuals who report either neuropathic pain or a reduced HRQoL score will be more closely examined, in order to identify CPSP or CRPS. Statistical analyses will be performed to determine whether haplotypes are associated with the development of either condition, and to determine the strength of this association.

ELIGIBILITY:
Inclusion Criteria:

* Provide written Informed Consent prior to participation in the study
* Be at lease 18, but not more than 80 years of age
* Have the ability to read and understand the study procedures and the use of the pain scales and have the ability to communicate meaningfully with the Study Investigator and staff.
* Be free of other physical, mental, or medical conditions, which, in the opinion of the Investigator, makes Study participation inadvisable
* Is scheduled to undergo open or arthroscopic shoulder surgery
* If the subject is a female of childbearing potential, have a negative pregnancy test on the day of surgery.

Exclusion Criteria:

- Has significant medical disease(s), laboratory abnormalities or conditions(s) that in the Investigator's judgment could compromise the Subject's welfare, ability to communicate with the Study staff, complete Study activities, or would otherwise contraindicate Study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing shoulder surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Scale | 6 months

SECONDARY OUTCOMES:
EQ-5D | 6 months
Numeric Rating Scale for pain | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hartrick, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - William Beaumont Hospitals, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan